CLINICAL TRIAL: NCT00052078
Title: Child/Adolescent Anxiety Multimodal Treatment Study
Brief Title: Child and Adolescent Anxiety Disorders (CAMS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U01MH064089 (NIH); U01MH064089 (NIH); DSIR 84-CTP
Record Dates: First submitted 2003-01-22; First posted 2003-01-23 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-08

CONDITIONS: Anxiety Disorders; Social Phobia; Generalized Anxiety Disorder
Keywords: Phobic Disorders; Anxiety, Separation
MeSH Terms: conditions — Anxiety Disorders; Phobia, Social; Generalized Anxiety Disorder; Phobic Disorders; Anxiety, Separation | interventions — Sertraline; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Sertraline (Active Comparator): Participants received sertraline for 12 weeks.
  Interventions: Drug: Sertraline (SRT)
- CBT (Active Comparator): Participants received cognitive behavioral therapy for 12 weeks
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- SRT + CBT (Active Comparator): Participants received both sertraline and CBT for 12 weeks.
  Interventions: Drug: Sertraline (SRT); Behavioral: Cognitive Behavioral Therapy (CBT)
- Placebo (Placebo Comparator): Participants received a placebo pill for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sertraline (SRT) — Participants were treated with sertraline.
  Other Names: Zoloft
  Arms: SRT + CBT; Sertraline
Behavioral: Cognitive Behavioral Therapy (CBT) — Participants received CBT.
  Arms: CBT; SRT + CBT
Drug: Placebo — Participants were treated with a placebo pill.
  Arms: Placebo

SUMMARY:
This randomized, controlled trial compared the efficacy of the medication sertraline (Zoloft®), cognitive-behavioral therapy, the combination of these treatments, and placebo for youth with anxiety disorders.

DETAILED DESCRIPTION:
Anxiety disorders are among the most common conditions affecting children and adolescents. These disorders impair school, social, and family functioning. When left untreated, they also put children at risk for major depression and substance abuse in late adolescence and adulthood. Previous studies demonstrated the efficacy of cognitive behavioral therapy and selective serotonin-reuptake inhibitors for the treatment of child anxiety disorders. This study is testing the relative and combined efficacy of cognitive behavioral therapy and selective serotonin reuptake inhibitors as compared to each other and pill placebo.

During Phase I of this two-phase study, 488 participants were randomly assigned to receive sertraline (Zoloft), cognitive behavioral therapy, a combination of these treatments, or a placebo for 12 weeks. Phase II involved a 6-month maintenance period for participants.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria for separation anxiety disorder, social phobia, or generalized anxiety disorder

Exclusion Criteria:

* Major neurological disorder or medical illness that would interfere with participation in the study

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 488 (Actual)
Dates: Start 2003-01; Primary Completion 2007-10 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - UCLA, Los Angeles, California
  - Johns Hopkins University, Baltimore, Maryland
  - NYSPI/Columbia University, New York, New York
  - Duke University, Durham, North Carolina
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburgh/WPIC, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Walkup JT, Albano AM, Piacentini J, Birmaher B, Compton SN, Sherrill JT, Ginsburg GS, Rynn MA, McCracken J, Waslick B, Iyengar S, March JS, Kendall PC. Cognitive behavioral therapy, sertraline, or a combination in childhood anxiety. N Engl J Med. 2008 Dec 25;359(26):2753-66. doi: 10.1056/NEJMoa0804633. Epub 2008 Oct 30. PMID 18974308
- [Result] Piacentini J, Bennett S, Compton SN, Kendall PC, Birmaher B, Albano AM, March J, Sherrill J, Sakolsky D, Ginsburg G, Rynn M, Bergman RL, Gosch E, Waslick B, Iyengar S, McCracken J, Walkup J. 24- and 36-week outcomes for the Child/Adolescent Anxiety Multimodal Study (CAMS). J Am Acad Child Adolesc Psychiatry. 2014 Mar;53(3):297-310. doi: 10.1016/j.jaac.2013.11.010. Epub 2013 Nov 28. PMID 24565357
- [Result] Ginsburg GS, Kendall PC, Sakolsky D, Compton SN, Piacentini J, Albano AM, Walkup JT, Sherrill J, Coffey KA, Rynn MA, Keeton CP, McCracken JT, Bergman L, Iyengar S, Birmaher B, March J. Remission after acute treatment in children and adolescents with anxiety disorders: findings from the CAMS. J Consult Clin Psychol. 2011 Dec;79(6):806-13. doi: 10.1037/a0025933. PMID 22122292
- [Result] Compton SN, Walkup JT, Albano AM, Piacentini JC, Birmaher B, Sherrill JT, Ginsburg GS, Rynn MA, McCracken JT, Waslick BD, Iyengar S, Kendall PC, March JS. Child/Adolescent Anxiety Multimodal Study (CAMS): rationale, design, and methods. Child Adolesc Psychiatry Ment Health. 2010 Jan 5;4:1. doi: 10.1186/1753-2000-4-1. PMID 20051130
- [Result] Compton SN, Peris TS, Almirall D, Birmaher B, Sherrill J, Kendall PC, March JS, Gosch EA, Ginsburg GS, Rynn MA, Piacentini JC, McCracken JT, Keeton CP, Suveg CM, Aschenbrand SG, Sakolsky D, Iyengar S, Walkup JT, Albano AM. Predictors and moderators of treatment response in childhood anxiety disorders: results from the CAMS trial. J Consult Clin Psychol. 2014 Apr;82(2):212-24. doi: 10.1037/a0035458. Epub 2014 Jan 13. PMID 24417601
- [Result] Kendall PC, Compton SN, Walkup JT, Birmaher B, Albano AM, Sherrill J, Ginsburg G, Rynn M, McCracken J, Gosch E, Keeton C, Bergman L, Sakolsky D, Suveg C, Iyengar S, March J, Piacentini J. Clinical characteristics of anxiety disordered youth. J Anxiety Disord. 2010 Apr;24(3):360-5. doi: 10.1016/j.janxdis.2010.01.009. Epub 2010 Feb 6. PMID 20206470
- [Derived] Strawn JR, Mills JA, Rothenberg R, Piacentini J, Peris TS, McCracken JT, Walkup JT. Initiation of Pharmacotherapy Following CBT in Anxious Youth: Results From the Child/Adolescent Anxiety Multimodal Study (CAMS). J Clin Psychiatry. 2022 Dec 5;84(1):22m14524. doi: 10.4088/JCP.22m14524. PMID 36479955
- [Derived] Crane ME, Norris LA, Frank HE, Klugman J, Ginsburg GS, Keeton C, Albano AM, Piacentini J, Peris TS, Compton SN, Sakolsky D, Birmaher B, Kendall PC. Impact of treatment improvement on long-term anxiety: Results from CAMS and CAMELS. J Consult Clin Psychol. 2021 Feb;89(2):126-133. doi: 10.1037/ccp0000523. PMID 33705168
- [Derived] Cervin M, Storch EA, Piacentini J, Birmaher B, Compton SN, Albano AM, Gosch E, Walkup JT, Kendall PC. Symptom-specific effects of cognitive-behavioral therapy, sertraline, and their combination in a large randomized controlled trial of pediatric anxiety disorders. J Child Psychol Psychiatry. 2020 Apr;61(4):492-502. doi: 10.1111/jcpp.13124. Epub 2019 Aug 30. PMID 31471911
- [Derived] Albano AM, Comer JS, Compton SN, Piacentini J, Kendall PC, Birmaher B, Walkup JT, Ginsburg GS, Rynn MA, McCracken J, Keeton C, Sakolsky DJ, Sherrill JT. Secondary Outcomes From the Child/Adolescent Anxiety Multimodal Study: Implications for Clinical Practice. Evid Based Pract Child Adolesc Ment Health. 2018;3(1):30-41. doi: 10.1080/23794925.2017.1399485. Epub 2017 Dec 5. PMID 30906874
- [Derived] Ginsburg GS, Becker-Haimes EM, Keeton C, Kendall PC, Iyengar S, Sakolsky D, Albano AM, Peris T, Compton SN, Piacentini J. Results From the Child/Adolescent Anxiety Multimodal Extended Long-Term Study (CAMELS): Primary Anxiety Outcomes. J Am Acad Child Adolesc Psychiatry. 2018 Jul;57(7):471-480. doi: 10.1016/j.jaac.2018.03.017. Epub 2018 May 9. PMID 29960692
- [Derived] Kiff CJ, Ernestus S, Gonzalez A, Kendall PC, Albano AM, Compton SN, Birmaher B, Ginsburg GS, Rynn M, Walkup JT, McCracken J, Piacentini J. The Interplay of Familial and Individual Risk in Predicting Clinical Improvements in Pediatric Anxiety Disorders. J Clin Child Adolesc Psychol. 2018;47(sup1):S542-S554. doi: 10.1080/15374416.2018.1460848. Epub 2018 Jun 7. PMID 29877727
- [Derived] Taylor JH, Lebowitz ER, Jakubovski E, Coughlin CG, Silverman WK, Bloch MH. Monotherapy Insufficient in Severe Anxiety? Predictors and Moderators in the Child/Adolescent Anxiety Multimodal Study. J Clin Child Adolesc Psychol. 2018 Mar-Apr;47(2):266-281. doi: 10.1080/15374416.2017.1371028. Epub 2017 Sep 28. PMID 28956620
- [Derived] Caporino NE, Sakolsky D, Brodman DM, McGuire JF, Piacentini J, Peris TS, Ginsburg GS, Walkup JT, Iyengar S, Kendall PC, Birmaher B. Establishing Clinical Cutoffs for Response and Remission on the Screen for Child Anxiety Related Emotional Disorders (SCARED). J Am Acad Child Adolesc Psychiatry. 2017 Aug;56(8):696-702. doi: 10.1016/j.jaac.2017.05.018. Epub 2017 Jun 6. PMID 28735699
- [Derived] Rynn MA, Walkup JT, Compton SN, Sakolsky DJ, Sherrill JT, Shen S, Kendall PC, McCracken J, Albano AM, Piacentini J, Riddle MA, Keeton C, Waslick B, Chrisman A, Iyengar S, March JS, Birmaher B. Child/Adolescent anxiety multimodal study: evaluating safety. J Am Acad Child Adolesc Psychiatry. 2015 Mar;54(3):180-90. doi: 10.1016/j.jaac.2014.12.015. Epub 2014 Dec 31. PMID 25721183
- [Derived] Gonzalez A, Peris TS, Vreeland A, Kiff CJ, Kendall PC, Compton SN, Albano AM, Birmaher B, Ginsburg GS, Keeton CP, March J, McCracken J, Rynn M, Sherrill J, Walkup JT, Piacentini J. Parental anxiety as a predictor of medication and CBT response for anxious youth. Child Psychiatry Hum Dev. 2015 Feb;46(1):84-93. doi: 10.1007/s10578-014-0454-6. PMID 24610431
- [Derived] Ginsburg GS, Becker EM, Keeton CP, Sakolsky D, Piacentini J, Albano AM, Compton SN, Iyengar S, Sullivan K, Caporino N, Peris T, Birmaher B, Rynn M, March J, Kendall PC. Naturalistic follow-up of youths treated for pediatric anxiety disorders. JAMA Psychiatry. 2014 Mar;71(3):310-8. doi: 10.1001/jamapsychiatry.2013.4186. PMID 24477837
- [Derived] Crawley SA, Caporino NE, Birmaher B, Ginsburg G, Piacentini J, Albano AM, Sherrill J, Sakolsky D, Compton SN, Rynn M, McCracken J, Gosch E, Keeton C, March J, Walkup JT, Kendall PC. Somatic complaints in anxious youth. Child Psychiatry Hum Dev. 2014 Aug;45(4):398-407. doi: 10.1007/s10578-013-0410-x. PMID 24129543

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 Setraline: Participants will receive sertraline for 12 weeks
  Sertraline: Participants will take sertraline for 12 weeks.
- 2 CBT: Participants will receive cognitive behavioral therapy for 12 weeks
  Cognitive Behavioral Therapy (CBT): Participants will receive CBT for 12 weeks.
- 3 Combination Setraline and CBT: Participants will receive a combination of sertraline and cognitive behavioral therapy for 12 weeks
  Sertraline: Participants will take sertraline for 12 weeks.
  Cognitive Behavioral Therapy (CBT): Participants will receive CBT for 12 weeks.
- 4 Placebo: Participants will receive placebo for 12 weeks
  Placebo: Participants will take placebo capsules for 12 weeks.
Period: Overall Study
Arm/Group | 1 Setraline | 2 CBT | 3 Combination Setraline and CBT | 4 Placebo
Started | 133 | 139 | 140 | 76
Completed | 110 | 133 | 127 | 61
Not Completed | 23 | 6 | 13 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Setraline | 2 CBT | 3 Combination Setraline and CBT | 4 Placebo | Total
Number analyzed (Participants) | 133 | 139 | 140 | 76 | 488
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 133 | 139 | 140 | 76 | 488
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 72 | 72 | 37 | 242
  Male | 72 | 67 | 68 | 39 | 246
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 1 | 0 | 6
  Asian | 4 | 1 | 6 | 1 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1 | 2
  Black or African American | 12 | 14 | 11 | 7 | 44
  White | 103 | 106 | 116 | 60 | 385
  More than one race | 12 | 15 | 5 | 7 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 133 | 139 | 140 | 76 | 488

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression - Improvement Scale
Description: The Clinical Global Impression - Improvement scale (CGI-I) is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention and rated as: 1-Very much improved; 2-Much improved; 3-Minimally improved; 4-No change; 5-Minimally worse; 6-Much worse; 7-Very much worse. Response rates are reported as a percentage of participants who score 1-Very much improved; 2-Much improved on the The Clinical Global Impression - Improvement scale.
Time Frame: Measured at Week 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 1 Setraline | 2 CBT | 3 Combination Setraline and CBT | 4 Placebo
Number analyzed (Participants) | 133 | 139 | 140 | 76
percentage of participants | 54.9 [46.4 to 63.1] | 59.7 [51.4 to 67.5] | 80.7 [73.3 to 86.4] | 23.7 [15.5 to 34.5]

ADVERSE EVENTS:
Groups:
- 3 Combination Setraline + CBT: Participants will receive a combination of sertraline and cognitive behavioral therapy for 12 weeks
  Sertraline: Participants will take sertraline for 12 weeks.
  Cognitive Behavioral Therapy (CBT): Participants will receive CBT for 12 weeks.
Arm/Group | 1 Setraline | 2 CBT | 3 Combination Setraline + CBT | 4 Placebo
Serious Adverse Events (participants affected / at risk) | 2/133 | 0/139 | 1/140 | 0/76
Other Adverse Events (participants affected / at risk) | 0/133 | 0/139 | 0/140 | 0/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Setraline (N=133) | 2 CBT (N=139) | 3 Combination Setraline + CBT (N=140) | 4 Placebo (N=76)
Worsening of Behavior (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — One participant in the sertraline group had a worsening of behavior that was attributed to the parents' increased limit setting on avoidance behavior; the event was considered to be possibly related to sertraline.
Oppositional-Defiant Behavior (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — One participant in the combination-therapy group had a worsening of preexisting oppositional-defiant behavior that resulted in psychiatric hospitalization; this event was considered to be unrelated to study treatment.
Tonsillectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — One participant in the sertraline group was medically hospitalized for a tonsillectomy. This event was considered unrelated to study treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No